CLINICAL TRIAL: NCT02551432
Title: Phase II Study of Pembrolizumab and Paclitaxel in Refractory Small Cell Lung Cancer
Brief Title: Pembrolizumab and Paclitaxel in Refractory Small Cell Lung Cancer
Acronym: MISP-MK3475
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Bhumsuk Keam, Clinical assistant professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MISP MK3475
Record Dates: First submitted 2015-07-07; First posted 2015-09-16 (Estimated); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Small Cell Lung Cancer
Keywords: pembrolizumab; paclitaxel
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — pembrolizumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paclitaxel pembrolizumab (Experimental): * PD-L1 Induction phase : Paclitaxel 175 mg/m2, Day 1 q 3weeks, intravenous,
  * Post Induction treatment phase: Paclitaxel 175 mg/m2, Day 1 q 3weeks (maximum up to total 6 cycles) + pembrolizumab 200 mg D1 q 3 weeks, intravenous,
  * Maintenance phase: pembrolizumab 200 mg D1 q 3 weeks, intravenous till PD or unacceptable toxicity
  Interventions: Drug: pembrolizumab, paclitaxel

INTERVENTIONS:
Drug: pembrolizumab, paclitaxel — pembrolizumab, paclitaxel
  Other Names: keytruda, taxol

SUMMARY:
Patients with refractory SCLC. Patients will be treated with paclitaxel and pembrolizumab.

DETAILED DESCRIPTION:
Open, uncontrolled, multi-center, phase II study.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be 20 years of age on day of signing informed consent.
3. Have measurable lesions based on RECIST 1.1.
4. Have provided tissue from an archival tissue sample obtained after the last previous treatment or newly obtained core or excisional biopsy of a tumor lesion.
5. Have a performance status of 0 or 1 on the ECOG Performance Scale.
6. Demonstrate adequate organ function as defined below 'adequate organ fuction laboratory values', all screening labs should be performed within 10 days of treatment initiation.

   'adequate organ fuction laboratory values' System Laboratory Value Hematological Absolute neutrophil count (ANC) ≥ 1,500 /mcL Platelets ≥100,000 / mcL Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L Renal Serum creatinine OR Measured or calculateda creatinine clearance (GFR can also be used in place of creatinine or CrCl)≤1.5 X upper limit of normal (ULN) OR ≥ 60 mL/min for subject with creatinine levels >1.5 X institutional ULN Hepatic Serum total bilirubin≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR
   * 5 X ULN for subjects with liver metastases Coagulation International Normalized Ratio (INR) or Prothrombin Time (PT)
   * 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants aCreatinine clearance should be calculated per institutional standard.
7. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
8. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 5.7.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
9. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has had a prior anti-cancer monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
4. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
5. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
6. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
7. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
8. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
9. Has an active infection requiring systemic therapy.
10. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
11. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
12. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
13. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
14. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
15. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected). (inactive HBsAg carriers with prophylactic antiviral agent are allowed)
16. Has received a live vaccine within 30 days prior to the first dose of trial treatment.
17. Has a known history of active TB (Bacillus Tuberculosis)
18. Has known hypersensitivity to MK-3475 or any of its excipients

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-09; Primary Completion 2017-12 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bhumsuk Keam, Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- Paclitaxel Pembrolizumab: * PD-L1 Induction phase : Paclitaxel 175 mg/m2, Day 1 q 3weeks, intravenous,
  * Post Induction treatment phase: Paclitaxel 175 mg/m2, Day 1 q 3weeks (maximum up to total 6 cycles) + pembrolizumab 200 mg D1 q 3 weeks, intravenous,
  * Maintenance phase: pembrolizumab 200 mg D1 q 3 weeks, intravenous till PD or unacceptable toxicity
  pembrolizumab, paclitaxel: pembrolizumab, paclitaxel
Period: Overall Study
Arm/Group | Paclitaxel Pembrolizumab
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Paclitaxel Pembrolizumab
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 17
Age, Continuous [Median (Full Range); unit: years] | 68.5 [54 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 26
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 26

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Tumor response will be assessed based on modified RECIST 1.1
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel Pembrolizumab
Number analyzed (Participants) | 26
Participants | 6

2. Secondary Outcome: Progression-free Survival
Description: Tumor response will be assessed based on modified RECIST 1.1
Time Frame: from first dose to disease progression or death due to any cause, whichever came first, up to 24months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel Pembrolizumab
Number analyzed (Participants) | 26
months | 5.0 [2.7 to 6.7]

3. Secondary Outcome: Overall Response (OS)
Description: Tumor response will be assessed based on modified RECIST 1.1
Time Frame: from first dose to death due to any cause, whichever came first, assessed up to 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel Pembrolizumab
Number analyzed (Participants) | 26
months | 9.1 [6.5 to 15.0]

4. Secondary Outcome: Safety(Toxicity)
Description: Safety will be assessed for all subjects and documented according to the CTCAE v4.0
Time Frame: 3 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: find out predictive biomarker for pembrolizumab. Factors potentially associated with pembrolizumab response will b analyzed for providing the rationale for future patient selection.
Time Frame: 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the first dose to 30 days after the last dose(till PD or unacceptable toxicity), an average of 1 year
Arm/Group | Paclitaxel Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 9/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel Pembrolizumab (N=26)
neutropenia (Blood and lymphatic system disorders) | 2
Pneumonia (Infections and infestations) | 2
type 1 Diabetes Mellitus (Endocrine disorders) | 1
febrile neutropenia (Blood and lymphatic system disorders) | 2
Asthenia (Musculoskeletal and connective tissue disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel Pembrolizumab (N=26)
anemia (Blood and lymphatic system disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 9
Anorexia (Gastrointestinal disorders) | 5
Nausea (Metabolism and nutrition disorders) | 4
Vomiting (Metabolism and nutrition disorders) | 2
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 6
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 5
Peripheral sensory neuropathy (Nervous system disorders) | 15
Hyponatremia (Blood and lymphatic system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-08): https://cdn.clinicaltrials.gov/large-docs/32/NCT02551432/Prot_SAP_000.pdf